CLINICAL TRIAL: NCT03056105
Title: The Psychobiological Effects of a One-Month Insight Meditation Retreat, a Sub-study of The Shamatha Project: A Longitudinal, Randomized Waitlist Control Study of Cognitive, Emotional, and Neural Effects of Intensive Meditation Training
Brief Title: The Psychobiological Effects of Participation in a One-Month Insight Meditation Retreat
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other); University of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: 230734
Record Dates: First submitted 2017-02-10; First posted 2017-02-17 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Aging
Keywords: Well-being, affiliation, inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, peripheral blood mononucleocytes, plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retreat: Participants registered for a one-month, residential Insight Meditation retreat held at Spirit Rock Meditation Center in either February or March, 2013
  Interventions: Other: Residential Insight Meditation Retreat
- Comparison: Experienced meditators from the Spirit Rock Meditation Community

INTERVENTIONS:
Other: Residential Insight Meditation Retreat — Retreats at Spirit Rock Meditation Center were led by teams of 6 experienced teachers. Participants practiced "noble silence"-refraining from eye contact as well as verbal and written communication-except during meetings with teachers. Teachers lead guided Insight meditation practices, as well as meditations on loving-kindness, compassion, empathetic joy, and equanimity. The daily schedule consisted of sitting and walking meditation sessions (30-45 mins) totaling 8-10 hours/day, meals, and short work meditations (sweeping, dishes, etc.). Seated meditation was practiced as a group in a meditation hall with approximately 80 participants. Walking meditation took place in adjoining halls or on the grounds. Participants lived on-site during the retreat and were provided with a vegetarian diet.
  Groups: Retreat

SUMMARY:
The purpose of this study was to examine how participation in a 1 month intensive Insight (vipassana) Meditation retreat (a) affects biological markers of cellular aging, social affiliation, and inflammation, which are important for physical health, longevity, and behavior, and (b) to relate observed biological changes to baseline levels and changes in psychological traits, which may underlie improvements in personal adaptive functioning.

DETAILED DESCRIPTION:
The investigators are specifically assessing the effects of retreat on telomere length and telomerase levels in participants' white blood cells, as well as plasma levels of interlukin-6 (IL-6), to assess how the retreat experience impacts these markers of cellular aging and inflammation. The hypotheses are that retreat participation will increase both telomere length and telomerase activity, but decrease IL-6 levels. The investigators will also assess the impact of retreat participation on oxytocin-a hormone involved in a number of physiological and behavioral processes, including affiliative bonds and stress responses-the hypothesis being that participation in the retreat will increase plasma oxytocin levels. The investigators will then explore how these and other biomarkers relate to psychological processes and personality traits, which may also be altered by participation in the meditation retreat.

ELIGIBILITY:
Inclusion Criteria:

* Previous meditation experience equivalent to two 5-10 day residential meditation retreats

Exclusion Criteria:

* Disclosure of potentially contagious blood-borne illness (e.g., HIV, Hepatitis, etc.) or other illnesses that might interfere with telomere or telomerase measurement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults with meditation experience
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-02-03 (Actual); Primary Completion 2014-02-04 (Actual); Study Completion 2014-02-04 (Actual)

PRIMARY OUTCOMES:
Telomerase | change from the start of retreat to three weeks into the retreat period
  an enzyme that repairs the shortening of telomeres that occurs during aging
Telomere length | change from the start of retreat to three weeks into the retreat period
  the repetitive sequence of DNA that serves as a protective cap to eukaryotic chromosomes, which protects from degradation and instability and is related to longevity
Interleukin-6 | change from the start of retreat to three weeks into the retreat period
  a primary measure of inflammation, which is influenced by psychological stress
Oxytocin | change from the start of retreat to three weeks into the retreat period
  an affiliative hormone associated with social bonding in both men and women, and which downregulates inflammatory cytokines

SECONDARY OUTCOMES:
Arginine Vasopressin | two measurements, three weeks apart
  a less commonly studied affiliative hormone also associated with close social bonds
Brain Derived Neurotrophic Factor | two measurements, three weeks apart
  a protein related to neuroplasticity, learning, and memory, which is decreased in depression
pro- and anti-inflammatory cytokines (IL-1b, IL-2, IL-4, IL-5, IL-10, IL-12 (p70), IL-13, IFN-γ, TNF-α) | two measurements, three weeks apart
  a family of proteins involved in generating and regulating the immune system
State-Trait Anxiety Inventory | two measurements, three weeks apart
  10 item scale designed to assess trait-anxiety (STAI; Spielberger et al., 1983)
Lifestyle Profile II | two measurements, three weeks apart
  Assesses health-promoting lifestyle factors (Walker et al., 1987)
Experience in Close Relationships, short form | two measurements, three weeks apart
  Assesses attachment anxiety (fear of rejection or abandonment) and avoidance (avoidance of intimacy and interdependence) (ECR-12: Lafontaine et al., 2015)
Mysticism Scale | two measurements, three weeks apart
  Assesses mystical experience and religious interpretation (M-Scale; Hood, 1975)
Non-attachment Scale | two measurements, three weeks apart
  Assesses non-attachment from a Buddhist perspective (NAS; Sahdra, Shaver & Brown, 2010)
Self-Assessed Wisdom Scale | two measurements, three weeks apart
  Assess five dimensions of wisdom: 1) Experience, 2) Emotional Regulation, 3) Reminiscence and Reflectiveness, 4) Openness, 5) Humor (SAWS; Webster, 2003)
Ego Resiliency Scale | two measurements, three weeks apart
  Assesses the ability to adapt one's level of control temporarily up or down as circumstances dictate (EGO; Block & Kremen, 1996)
Five Facet Mindfulness Questionnaire | two measurements, three weeks apart
  Assesses five facets of mindfulness: 1) Non-reactivity to Inner Experience, 2) Observing 3) Acting with Awareness, 4) Describing, and 5) Non-judging of Experience (FFMQ; Baer et al., 2006)
Center for Epidemiological Studies Depression Scale | two measurements, three weeks apart
  Assesses depressive symptomatology (CES-D; Radloff, 1977)
Psychological Wellbeing Scale | two measurements, three weeks apart
  Assess autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance (PWBS; Ryff, 1989)
Three Dimensional Wisdom Scale | two measurements, three weeks
  Assess three dimensions of wisdom: 1) Cognitive, 2) Reflective, and 3) Affective (3-DWS; Ardelt, 2003)
Big Five Inventory | two measurements, three weeks
  Assesses extraversion, agreeableness, conscientiousness, openness to experience, neuroticism (BFI; Goldberg, 1993)
Difficulties in Emotion Regulation Scale | two measurements, three weeks
  Assesses non-acceptance to one's emotional responses, difficulty achieving goals, impulsiveness, lack of emotional awareness, access to emotion regulation strategies, emotional clarity (DERS; Gratz & Roemer, 2004)

OTHER OUTCOMES:
Gene Expression of genes relating to inflammation and telomere regulation | two measurements, three weeks
  PBMC RNA for exploratory gene expression studies

CONTACTS AND LOCATIONS:
Overall Officials: Clifford D Saron, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Conklin QA, King BG, Zanesco AP, Lin J, Hamidi AB, Pokorny JJ, Alvarez-Lopez MJ, Cosin-Tomas M, Huang C, Kaliman P, Epel ES, Saron CD. Insight meditation and telomere biology: The effects of intensive retreat and the moderating role of personality. Brain Behav Immun. 2018 May;70:233-245. doi: 10.1016/j.bbi.2018.03.003. Epub 2018 Mar 5. PMID 29518528